CLINICAL TRIAL: NCT01045083
Title: Randomized, Observer-blind, Placebo-controlled, Four-way Cross-over Study to Study the Ability of Functional Magnetic Resonance Imaging (fMRI) of the Brain to Detect and Characterize the Effects of Single Doses of a Selective Serotonin Reuptake Inhibitor (Escitalopram [Lexapro]), a Dopamine
Brief Title: A Study of the Ability of Functional Magnetic Resonance Imaging (fMRI) to Detect and Characterize the Effects of Two Marketed Centrally Active Drugs, Placebo, and RO4917523 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: BP22651
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine; Escitalopram; Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RO4917523; Drug: escitalopram; Drug: methylphenidate; Drug: placebo

INTERVENTIONS:
Drug: RO4917523 — Oral single dose
Drug: escitalopram — Oral single dose
  Other Names: Lexapro
Drug: methylphenidate — Oral single dose
  Other Names: Ritalin
Drug: placebo — Oral single dose

SUMMARY:
This is an exploratory study to evaluate the usefulness of fMRI as a biomarker to characterize the response to three centrally active drugs and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 45 years of age
* In good general health
* Weight of ≥120 lbs (55 kg) and a body mass index (BMI) between 18 to 30kg/m²
* Males and females with reproductive potential: willing to use a reliable method of contraception

Exclusion Criteria:

* Evidence of clinically significant disease
* Medical or surgical condition that could alter the absorption, metabolism, or elimination of drugs
* Family history of sudden death or ventricular arrhythmia
* History of any psychiatric disorder and/or marked anxiety
* History of glaucoma
* History (including family) of motor tic or diagnosis of Tourette's syndrome
* Active suicide ideation
* Contraindication to MRI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of fMRI to detect and characterize the effect of the three drugs on brain activity at rest and during emotional stimuli | 8 weeks

SECONDARY OUTCOMES:
To evaluate the ability of other behavioural paradigms/scales to detect drug effects | 8 weeks
To correlate the fMRI measures with the clinical/behavioral measures | 8 weeks
To investigate the safety of single doses of RO4917523 in healthy volunteers | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- La Jolla, California, United States